CLINICAL TRIAL: NCT01280747
Title: Examination of Pregabalin Access for Treatment of Indicated Pain Disorders: the ExPAND Study
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081247
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2012-06

CONDITIONS: Fibromyalgia; Painful Diabetic Peripheral Neuropathy
Keywords: Prior authorization; Fibromyalgia; Painful Diabetic Peripheral Neuropathy; Policy; Real World Data
MeSH Terms: conditions — Fibromyalgia | interventions — Prior Authorization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Eligible fibromyalgia patients receive usual care with pregabalin prior authorization requirements in place
  Interventions: Other: prior authorization
- 2: Eligible fibromyalgia patients receive usual care without pregabalin prior authorization requirements in place
  Interventions: Other: no prior authorization
- 3: Eligible painful diabetic peripheral neuropathy patients receive usual care with pregabalin prior authorization requirements in place
  Interventions: Other: prior authorization
- 4: Eligible painful diabetic peripheral neuropathy patients receive usual care without pregabalin prior authorization requirements in place
  Interventions: Other: no prior authorization

INTERVENTIONS:
Other: prior authorization — This is a naturalistic study. The physician will prescribe medication(s) as appropriate
  Groups: 1
Other: no prior authorization — This is a naturalistic study. The physician will prescribe medication(s) as appropriate
  Groups: 2
Other: prior authorization — This is a naturalistic study. The physician will prescribe medication(s) as appropriate
  Groups: 3
Other: no prior authorization — This is a naturalistic study. The physician will prescribe medication(s) as appropriate
  Groups: 4

SUMMARY:
The investigators hypothesize that fibromyalgia (FM) and painful diabetic peripheral neuropathy (pDPN) patients with access restrictions on pregabalin will lead to higher healthcare resource use and cost compared to patients without such restrictions on pregabalin in a naturalistic setting. The randomization will occur at the physician level and not the patient level.

DETAILED DESCRIPTION:
This trial was terminated prematurely on April 2, 2012, due to the inability to recruit the planned number of subjects. The decision to terminate the trial was not based on any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* A physician-confirmed diagnosis of either pDPN or FM, but not both.
* Initiation of a medication for pDPN or FM is clinically indicated, either as monotherapy or in combination with other treatments, as determined by the treating physician, and agreed to by the patient.
* No prior pregabalin use or pregabalin PA requests.

Exclusion Criteria:

* Age < 18 years at time of study enrollment.
* Females or are partners of males currently pregnant/lactating or intending to become pregnant in the next 6 months
* Physician-confirmed diagnosis of both pDPN and FM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are six practice types that are expected to be able to provide patients to this study. Of these, four (internal medicine, family/general practitioners, neurologists, and anesthesia/pain physicians) will be expected to enroll patients into both pDPN and FM disease groups. The fifth group, rheumatology physicians, will be expected to enroll patients into the FM cohort only and the sixth group, endocrinologists, will be expected to enroll patients into the pDPN cohort only.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Quantify the between-group difference (baseline to 6 mo.) in direct all-cause medical costs for patients with pDPN and FM in real-world treatment settings with a prior authorization (PA) versus no PA policy in place restricting access to | 6 months
pregabalin | 6 months
Evaluate the within-group differences (baseline to 6 mo.) in pain alleviation (using the 11 point numerical rating scale) in patients with pDPN and FM in real-world settings with a PA versus no PA policy in place restricting access to | 6 months
pregabalin. | 6 months

SECONDARY OUTCOMES:
Describe how pharmacologic treatment patterns for pDPN or FM differ between groups with PA and without PA in patients being treated in a naturalistic outpatient care setting, and who are followed for 6 mo. | 6 months
Describe non-pharmacologic treatment patterns in pDPN and FM patients in groups with PA versus no PA while being treated in a naturalistic outpatient care setting, and who are followed for 6 mo. | 6 months
Subset of patients who have at least 6 mo. pre-study time in the HIRD (HealthCore Integrated Research DatabaseSM) a within-group costs analysis (all cause) comparing pre-study healthcare utilization costs for the 6 mo. pre-baseline with on-study | 6 months
healthcare utilization costs (baseline to 6 mo.). | 6 months
Assess changes (baseline through 6 mo.) in other PRO measures in pDPN and FM patients subject to PA requirements for pregabalin versus those with no PA. | 6 months
Compare the within-group differences (baseline to 6 mo.) in pain alleviation (using the NRS-11 scale) between groups (PA versus no PA), by condition (pDPN or FM). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (17):
  - Osteoporosis Medical Center, Beverly Hills, California
  - Torrence Clinical Research, Lomita, California
  - Joo-Hyung Lee, MD, Orange, California
  - Thomas M Dawes Jr. MD, Santa Maria, California
  - Tulare Family Practice Medical Group, Tulare, California
  - Affiliates of Medical Specialties, West Hills, California
  - Primary Care Specialists LLC, Atlanta, Georgia
  - Southern Family Medical Center, PC, Augusta, Georgia
  - WeCareMD, P.C., Hiram, Georgia
  - Pain Care LLC, Stockbridge, Georgia
  - Broadway Family Medicine, Anderson, Indiana
  - Duneland Health and Wellness Institute, Chesterton, Indiana
  - Alan S. Goldenhar, DPM, No Conway, New Hampshire
  - Endocrine Associates of Long Island, P.C., Smithtown, New York
  - Mound Family Practice, Miamisburg, Ohio
  - Piqua Family Practice, Piqua, Ohio
  - Ettrick Health Center, Ettrick, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081247&StudyName=Examination%20of%20Pregabalin%20Access%20for%20Treatment%20of%20Indicated%20Pain%20Disorders%3A%20the%20ExPAND%20Study%20